CLINICAL TRIAL: NCT02122029
Title: A Nine-Year Follow-up of Intensive Lifestyle Intervention vs Surgery to Treat Morbidly Obese Women: a Non-randomized Human Subject Research.
Brief Title: Lifestyle vs.Surgery for Morbid Obesity Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Principal Investigator, M. Yannakoulia, Associate Professor, Harokopio University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVS
Record Dates: First submitted 2014-04-15; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Morbid Obesity
Keywords: Lifestyle intervention; Bariatric surgery; Weight management; Physical activity
MeSH Terms: conditions — Obesity, Morbid; Motor Activity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bariatric Surgery (Experimental)
  Interventions: Behavioral: Lifestyle counselling
- Lifestyle counselling (Experimental)
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Behavioral: Lifestyle counselling — Behavioral techniques for weight management
  Arms: Bariatric Surgery
Procedure: Bariatric Surgery — Vertical Banding Gastroplasty
  Arms: Lifestyle counselling

SUMMARY:
The purpose of the current study is to determine whether an intensive lifestyle intervention was as effective as surgery to treat morbid obesity nine years post-intervention.

DETAILED DESCRIPTION:
Behavioral/lifestyle interventions produce acceptable success in treating moderately obese subjects. However, their effectiveness on weight loss and maintenance in morbidly obese subjects remains elusive.

Twenty-nine morbidly obese females participated in this non-randomized study. Fifteen subjects were assigned to the lifestyle group and 14 underwent vertical banded gastroplasty. Subjects in the lifestyle group attended 30 behavioral modification sessions over three years, whereas the surgery group received the standard of care nutrition. Body weight, resting metabolic rate, physical activity, body composition measurements and dietary intake data were assessed at standard time points during the first 3 years post-intervention. Follow-up data on body weight and physical activity were also collected 9 years later.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* Age ≥ 18 years
* BMI ≥ 40 kg/m2
* Absence of mental illness as determined by evaluation by an experienced psychiatrist
* Additional inclusion criteria for vertical banded gastroplasty were history of multiple, non-successful, previous attempts for weight loss

Ages: 21 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2003-02; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The weight lost (kg) and maintained (kg) following each intervention (bariatric surgery and behavioural modification) | 9 years

SECONDARY OUTCOMES:
Physical Activity Level post bariatric surgery and behavioural modification of morbid obese patients. | 9 years
Resting Metabolic Rate (kcal/d) post bariatric surgery and behavioral modofication in morbid obese patients. | 3 years
Fat mass (kg) and fat free mass (kg) post bariatric surgery and behavioural modification in morbid obese patients. | 3 years
Changes in dietary intake and eating habits post bariatric surgery and behavioural modification. | 3 years
  Dietary intake measured as energy intake (kcal/d) derived from fat, protein and carbohydrate.
  Eating habits were reflected by the reported consumption of fruits, vegetables, sweets (portions/d).

CONTACTS AND LOCATIONS:
Overall Officials: Labros S Sidossis, Professor, Study Director — Department of Internal Medicine, Surgery, and Nutrition and Metabolism, University of Texas Medical Branch at Galveston, Texas, USA
Locations (1):
- Harokopio University, Athens, Greece